CLINICAL TRIAL: NCT00594529
Title: Feasibility Study of Neoadjuvant Chemotherapy Modified FOLFOX6 for Resectable Liver Metastases of Colorectal Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyoto University (Other)
Responsible Party: Dept. Surgery, Kyoto Univ., Dept. Surgery, Kyoto Univ.
Organization: Kyoto University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-206; UMIN000000961
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-08

CONDITIONS: Colorectal Cancer; Liver Metastasis
Keywords: Neoadjuvant chemotherapy; Metastatic liver lesions from colorectal cancers
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surgical Procedures, Operative

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Liver resection for metastatic liver lesions

SUMMARY:
The purpose of this study is to evaluate the safety of liver resection for metastatic, resectable lesions from colorectal cancers after systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed as colorectal adenocarcinomas, including cecal, appendiceal, and anal canal cancers.
2. Liver lesions are measurable by spiral CT or SPIO-MRI scans.
3. Extrahepatic lesions include lung metastases which can be resected curatively.
4. Curative resection for metastatic lesions can be performed with residual hepatic functions preserved.
5. No prior treatment histories for liver lesions, including L-OHP regimens, hepatectomy, hepatic arterial infusion, MCT, or RFA
6. No evidence of chronic hepatic diseases which affect systemic chemotherapy and/or surgical resection
7. Performance status (ECOG): 0-1
8. Vital organ functions, including hematopoietic, cardiac, respiratory and renal functions, are preserved.

Exclusion Criteria:

Excluded are cases with conditions as below:

1. Peritoneal or pleural fluid retention to be drained.
2. Multiple malignancies to be treated.
3. Peripheral neural disturbances.
4. Active infectious diseases.
5. Severe watery diarrhea.
6. Mental disturbances.
7. Treatment history of continuous, oral or intravenous steroid therapy.
8. Previous history of ischemic heart diseases.
9. Coexistent severe diseases including pulmonary fibrosis, interstitial pneumonia, ileus, uncontrollable diabetes, cardiac dysfunction, hepatic failure, or renal failure.
10. Pregnant.
11. Previous history of severe drug-induced allergy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Curative resection rates of liver metastases | 2 years after the operations

SECONDARY OUTCOMES:
Completion rates of neoadjuvant chemotherapy | 2 years after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoto University Hospital, Kyoto, Japan

REFERENCES:
- [Derived] Nagayama S, Hasegawa S, Hida K, Kawada K, Hatano E, Nakamura K, Seo S, Taura K, Yasuchika K, Matsuo T, Zaima M, Kanazawa A, Terajima H, Tada M, Adachi Y, Nishitai R, Manaka D, Yoshimura T, Doi K, Horimatsu T, Mitsuyoshi A, Yoshimura K, Niimi M, Matsumoto S, Sakai Y, Uemoto S. Multi-institutional phase II study on the feasibility of liver resection following preoperative mFOLFOX6 therapy for resectable liver metastases from colorectal cancers. Int J Clin Oncol. 2017 Apr;22(2):316-323. doi: 10.1007/s10147-016-1050-5. Epub 2016 Oct 17. PMID 27752787